CLINICAL TRIAL: NCT01118273
Title: A Double-Blind, Randomized, Pilot Study Assessing the Analgesic and Hypnotic Effect of Naproxen Sodium and Diphenhydramine Combination in Dental Pain
Brief Title: Evaluate Analgesic/Sedative Efficacy of Naproxen Sodium and Diphenhydramine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13053
Record Dates: First submitted 2010-04-15; First posted 2010-05-06 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Sleep
Keywords: Naproxen sodium; Diphenhydramine; Drugs, Investigational
MeSH Terms: interventions — Naproxen; Ibuprofen; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg (Experimental)
  Interventions: Drug: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg
- Naproxen Sodium 440 mg (BAYH6689) (Active Comparator)
  Interventions: Drug: Naproxen Sodium 440 mg (BAYH6689)
- Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg (Experimental)
  Interventions: Drug: Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg
- Naproxen Sodium 220 mg (BAYH6689) (Active Comparator)
  Interventions: Drug: Naproxen Sodium 220 mg (BAYH6689)
- DPH 50mg (Active Comparator)
  Interventions: Drug: DPH 50mg
- Ibuprofen 400 mg / Diphenhydramine citrate 76 mg (Active Comparator)
  Interventions: Drug: Ibuprofen 400 mg / Diphenhydramine citrate 76 mg

INTERVENTIONS:
Drug: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg — Participants received 2 tablets of Naproxen Sodium 220 mg and 2 tablets of Diphenhydramine hydrochloride (DPH) 25 mg, single dose, orally.
  Arms: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg
Drug: Naproxen Sodium 440 mg (BAYH6689) — Participants received 2 tablets of Naproxen Sodium 220mg and 2 tablets of placebo, single dose, orally.
  Arms: Naproxen Sodium 440 mg (BAYH6689)
Drug: Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg — One dose of naproxen sodium 220 mg plus diphenhydramine 50 mg
  Arms: Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg
Drug: Naproxen Sodium 220 mg (BAYH6689) — Participants received 1 tablet of Naproxen Sodium 220 mg and 3 tablets of placebo, single dose, orally.
  Arms: Naproxen Sodium 220 mg (BAYH6689)
Drug: DPH 50mg — Participants received 2 tablets of Diphenhydramine hydrochloride (DPH) 25 mg and 2 tablets of placebo, single dose, orally.
  Arms: DPH 50mg
Drug: Ibuprofen 400 mg / Diphenhydramine citrate 76 mg — Participants received 2 tablets of Advil PM (ibuprofen 200 mg and diphenhydramine citrate 38 mg) and 2 tablets of Placebo, single dose, orally.
  Arms: Ibuprofen 400 mg / Diphenhydramine citrate 76 mg

SUMMARY:
The objectives of the study are to evaluate the analgesic and hypnotic efficacy of naproxen sodium and diphenhydramine combination when compared to naproxen sodium, diphenhydramine, and an ibuprofen and diphenhydramine combination

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers between 16-45 years of age;
* Scheduled to undergo surgical removal of 1 to 3 impacted third molars, one of which must be at least a partial bony mandibular impaction;
* Have moderate to severe postoperative pain on the Categorical Pain Rating Scale and a score of >/= 50 mm on the 100-mm visual analog Pain Severity Rating Scale by 2030 h +/- 15 minutes on the day of surgery;
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g. oral or patch contraceptives, intrauterine device, Depo-Provera, or double-barrier and have a negative pregnancy test at Screening and prior to surgery. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy;
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial, (subjects <18 years of age must sign a written assent and have parental or guardian consent).

Exclusion Criteria:

* History of hypersensitivity to naproxen, diphenhydramine, nonsteroidal antiinflammatory drugs (NSAIDS), tramadol, aspirin or any other antihistamine and similar pharmacological agents or components of the products;
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years;
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than 50 percent obstruction (polyposis nasi, marked septal deviation) that can interfere with the conduct of the study in the judgment of the investigator;
* Current or past history of bleeding disorder(s);
* Acute illness or local infection prior to surgery that can interfere with the conduct of the study in the judgment of the investigator;
* Chronic use of antihistamines defined as using 5 or more times a week for 2 or more consecutive weeks during the past 3 months;
* Positive alcohol breathalyzer test and negative urine drug test prior to surgery;
* Females who are pregnant or lactating;
* Chronic or severe sleep problems that do not respond to Over the counter (OTC) medication and requires a prescription hypnotic or sedative;

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 162 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg: Participants received 1 tablet of Naproxen Sodium 220 mg and 2 tablets of Diphenhydramine hydrochloride (DPH) 25 mg and 1 tablet of placebo, single dose, orally.
Period: Overall Study
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Started | 27 | 27 | 27 | 27 | 27 | 27
Completed | 27 | 27 | 27 | 27 | 27 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg | Naproxen Sodium 440 mg (BAYH6689) | Total
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (2.8) | 20 (2.8) | 19 (2.0) | 19 (3.0) | 19 (2.5) | 20 (2.6) | 19 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 10 | 19 | 12 | 12 | 84
  Male | 11 | 12 | 17 | 8 | 15 | 15 | 78
Baseline Categorical Pain Rating Scale [Number; unit: Participants]
  No pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mild pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate pain | 15 | 14 | 14 | 17 | 21 | 14 | 95
  Severe pain | 12 | 13 | 13 | 10 | 6 | 13 | 67

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time Measured by Actigraphy
Description: Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects. In calculating the total sleep time, subjects who took rescue medication were treated as "awake" from the time the rescue medication was given until the end of the sleep period. In addition, if subjects rescued before sleep onset, their total sleep time was set to zero.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Minutes | 339.80 [259 to 420] | 304.60 [224 to 385] | 413.89 [333 to 494] | 308.89 [228 to 389] | 76.35 [-4 to 157] | 335.68 [254 to 417]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.54, ANCOVA

2. Secondary Outcome: Wake After Sleep Onset (WASO) Measured by Actigraphy
Description: Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects. WASO was defined as minutes of awake during the period of sleep onset and offset, where sleep onset is the first 20-minute block with 19 minutes of sleep.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Minutes | 139.96 [70 to 210] | 190.91 [121 to 261] | 75.66 [7 to 144] | 145.67 [72 to 219] | 428.34 [351 to 506] | 129.02 [59 to 199]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.31, ANCOVA

3. Secondary Outcome: Sleep Latency Measured by Actigraphy
Description: Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects. Sleep latency was defined as minutes to sleep onset since dosing, where sleep onset was the first 20-minute block with 19 minutes of sleep. For subjects who had not achieved sleep onset (e.g., due to taking rescue medication before achieving sleep onset), sleep latency was considered as censored at the time of wakening.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Minutes | 29.17 [9 to 50] | 32.81 [12 to 53] | 46.77 [27 to 67] | 31.58 [10 to 53] | 41.05 [18 to 64] | 36.38 [16 to 57]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.45, Log Rank

4. Secondary Outcome: Global Assessment of Study Medication as a Sleep-aid
Description: Subject rating of following question with 0 being poor to 4 being excellent: How would you rate the study medication you received as a sleep aid?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  Poor | 1 | 6 | 2 | 4 | 6 | 0
  Fair | 4 | 4 | 3 | 6 | 7 | 6
  Good | 8 | 7 | 7 | 6 | 3 | 9
  Very good | 5 | 4 | 8 | 3 | 2 | 7
  Excellent | 4 | 1 | 3 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Karolinska Sleep Diary - Sleep Quality
Description: Subject rating of following question with 1 being very poor and 5 being very good: How was your sleep?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  1 = Very poor | 1 | 4 | 1 | 1 | 1 | 0
  2 = Rather poor | 2 | 0 | 2 | 2 | 5 | 1
  3 = Neither poor nor good | 6 | 11 | 3 | 7 | 3 | 10
  4 = Rather good | 11 | 5 | 14 | 9 | 9 | 9
  5 = Very good | 2 | 2 | 3 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.05, ANCOVA

6. Secondary Outcome: Karolinska Sleep Diary - Calmness of Sleep
Description: Subject rating of following question with 1 being very restless and 5 being very calm: How calm was your sleep?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  1 = Very restless | 0 | 2 | 1 | 1 | 1 | 0
  2 = Rather restless | 1 | 7 | 6 | 5 | 7 | 7
  3 = Neither restless nor calm | 5 | 4 | 3 | 7 | 3 | 5
  4 = Rather calm | 16 | 6 | 12 | 6 | 6 | 8
  5 = Very calm | 0 | 3 | 1 | 1 | 1 | 2
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.019, ANCOVA

7. Secondary Outcome: Karolinska Sleep Diary - Easiness to Fall Asleep
Description: Subject rating of following question with 1 being very difficult to 5 being very easy: How easy was it to fall asleep?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  1 = Very difficult | 0 | 5 | 1 | 3 | 1 | 0
  2 = Rather difficult | 3 | 3 | 2 | 5 | 6 | 5
  3 = Neither difficult nor easy | 10 | 11 | 11 | 3 | 7 | 7
  4 = Rather easy | 8 | 2 | 8 | 7 | 4 | 9
  5 = Very easy | 1 | 1 | 1 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.018, ANCOVA

8. Secondary Outcome: Karolinska Sleep Diary - Premature Awakening
Description: Subject rating of following question with 1 being woke up much too early to 3 being no: Premature awakening?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  1 = Woke up much too early | 5 | 6 | 2 | 6 | 8 | 5
  2 = Woke up somewhat too early | 8 | 10 | 12 | 7 | 6 | 13
  3 = No | 9 | 6 | 9 | 7 | 4 | 4
Statistical Analysis 1: Comparison: Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.03, Cochran-Mantel-Haenszel

9. Secondary Outcome: Karolinska Sleep Diary - Ease of Awakening
Description: Subject rating of following question with 1 being very difficult to 5 being very easy: Ease of awakening?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  1 = Very difficult | 0 | 1 | 0 | 1 | 0 | 0
  2 = Rather difficult | 1 | 0 | 2 | 1 | 1 | 0
  3 = Neither difficult nor easy | 1 | 7 | 5 | 1 | 3 | 4
  4 = Rather easy | 15 | 8 | 8 | 15 | 9 | 14
  5 = Very easy | 5 | 6 | 8 | 2 | 5 | 4
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.76, Cochran-Mantel-Haenszel

10. Secondary Outcome: Karolinska Sleep Diary - Well Rested
Description: Subject rating of following question with 1 being not rested at all to 3 being completely rested: Well-rested?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  1 = Not rested at all | 1 | 4 | 0 | 0 | 3 | 1
  2 = Somewhat unrested | 13 | 14 | 14 | 12 | 14 | 17
  3 = Completely rested | 8 | 4 | 9 | 8 | 1 | 4
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.015, ANCOVA

11. Secondary Outcome: Karolinska Sleep Diary - Sufficient Sleep
Description: Subject rating of following question with 1 being no, definitely too little to 5 being yes, definitely enough: Did you get enough (sufficient) sleep?
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 22 | 22 | 23 | 20 | 18 | 22
Participants
  1 = No, definitely too little | 1 | 4 | 0 | 1 | 2 | 1
  2 = No, much too little | 4 | 3 | 2 | 1 | 4 | 1
  3 = No, somewhat too little | 4 | 4 | 3 | 4 | 8 | 6
  4 = Yes, almost enough | 10 | 8 | 14 | 10 | 4 | 12
  5 = Yes, definitely enough | 3 | 3 | 4 | 4 | 0 | 2
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.04, Cochran-Mantel-Haenszel

12. Secondary Outcome: Total Sleep Time by Subject Assessment
Description: Subject responded to: Please estimate the number of hours and minutes you think that you slept.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Minutes | 306.32 [231 to 381] | 309.97 [235 to 385] | 339.08 [264 to 414] | 309.23 [234 to 384] | 160.49 [85 to 236] | 299.58 [223 to 376]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.95, ANCOVA

13. Secondary Outcome: Sleep Quality Index
Description: Sleep Quality Index is the mean score of items, 'sleep quality', 'calm sleep', 'ease falling asleep', and 'slept throughout' on the Karolinska Sleep Diary, ranges from 1 (worst possible) to 5 (best possible).
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population with available data (missing values were not imputed).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Scores on a scale | 3.49 [3.1 to 3.9] | 2.89 [2.5 to 3.3] | 3.40 [3.0 to 3.8] | 3.12 [2.7 to 3.5] | 2.96 [2.6 to 3.4] | 3.37 [3.0 to 3.7]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.05, Cochran-Mantel-Haenszel

14. Secondary Outcome: Overall Rating of Severity in Categorical Pain Rating Scale Score
Description: Subject responded to question, 'My pain at this time is' by selecting one of the following choices: no pain (0), mild pain (1), moderate pain (2), or severe pain (3).
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Scores on a scale
  Baseline | 2.44 (0.51) | 2.48 (0.51) | 2.48 (0.51) | 2.48 (0.51) | 2.37 (0.49) | 2.22 (0.42)
  Post-Baseline | 1.26 (1.02) | 1.48 (1.05) | 1.26 (0.94) | 1.78 (0.97) | 2.67 (0.62) | 1.41 (1.01)

15. Secondary Outcome: Change From Baseline in Categorical Pain Rating Scale Score
Description: Subjects responded to question, 'My pain at this time is' with following choices: no pain (0), mild pain (1), moderate pain (2), or severe pain (3). Subjects completed this question at baseline (post-dental surgery) and after sleep period. The following measure is the change in pain rating from baseline.
Time Frame: Baseline and up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Scores on a scale | -1.2 [-1.5 to -0.8] | -1.0 [-1.3 to -0.6] | -1.2 [-1.5 to -0.8] | -0.7 [-1.0 to -0.3] | 0.3 [-0.1 to 0.6] | -0.9 [-1.3 to -0.6]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.42, ANCOVA

16. Secondary Outcome: Overall Rating of Severity in Visual Analog Scale (VAS) Score
Description: Subjects marked a line on a 100-mm scale to indicate the severity of pain they are experiencing from 0 being no pain to 100 being worse possible pain.
Time Frame: At 10 hours
Population: ITT (Intent to Treat) Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Scores on a scale
  Baseline | 76.11 (11.6) | 77.26 (13.1) | 78.19 (13.4) | 73.70 (12.3) | 79.15 (9.76) | 73.11 (10.5)
  Post-Baseline | 32.11 (31.1) | 40.30 (33.0) | 30.33 (28.6) | 48.59 (33.4) | 84.26 (19.9) | 38.19 (32.9)
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg; Test type: Superiority or Other; p = 0.35, ANCOVA

17. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Score
Description: Subjects completed the VAS scale at baseline (post-dental surgery) and after completion of the sleep period. Subjects marked a line on a 100-mm scale to indicate the severity of pain they are experiencing from 0 being no pain to 100 being worse possible pain.This measure indicates the change in pain severity rating on the VAS scale from baseline.
Time Frame: Baseline and up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Scores on a scale | -44.04 [-55.1 to -33.0] | -36.65 [-47.7 to -25.6] | -47.26 [-58.4 to -36.2] | -25.89 [-37.0 to -14.8] | 6.00 [-5.1 to 17.1] | -35.89 [-47.0 to -24.8]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.35, ANCOVA

18. Secondary Outcome: Overall Rating of Pain Relief
Description: Subjects responded to question, "Overall, the relief from my starting pain was" by checking one of the following choices: no relief (0), a little relief (1), some relief (2), a lot of relief (3), complete relief (4).
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Participants
  No relief | 1 | 3 | 2 | 6 | 11 | 4
  A little relief | 4 | 4 | 3 | 3 | 9 | 2
  Some relief | 8 | 7 | 5 | 4 | 5 | 5
  A lot relief | 12 | 10 | 13 | 11 | 2 | 13
  Complete relief | 2 | 3 | 4 | 3 | 0 | 3
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.72, ANCOVA

19. Secondary Outcome: Time to Rescue Medication
Description: Subjects were allowed to "rescue" and take a non-study pain reliever if the pain was not tolerable. This measure represents for the time to taking rescue medication from the time the subject took study treatment.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Minutes | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | NA [NA to NA] — Technically the data is not computable due to insufficient number of events | NA [NA to NA] — Technically the data is not computable due to insufficient number of events
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs DPH 50mg; Test type: Superiority or Other; p = 0.001, Log Rank

20. Secondary Outcome: Cumulative Proportion of Participants Taking Rescue Medication by Hour
Description: Subjects were allowed to "rescue" and take a non-study pain reliever if the pain was not tolerable. This measure represents for the proportion of subjects who rescued in the study.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Participants
  1 hour | 2 | 3 | 0 | 1 | 4 | 0
  2 hours | 6 | 9 | 5 | 9 | 17 | 7
  3 hours | 8 | 11 | 5 | 9 | 20 | 7
  4 hours | 10 | 11 | 5 | 10 | 21 | 7
  5 hours | 11 | 11 | 5 | 11 | 24 | 7
  6 hours | 11 | 11 | 6 | 12 | 25 | 9
  7 hours | 11 | 12 | 7 | 13 | 25 | 10
  8 hours | 11 | 12 | 7 | 13 | 25 | 10
  9 hours | 11 | 12 | 8 | 13 | 25 | 11
  10 hours | 12 | 12 | 8 | 13 | 25 | 11

21. Secondary Outcome: Global Assessment of Study Medication as a Pain Reliever
Description: Subject responded to question, 'How would you rating this study medication you received as a pain-reliever?' with the following choices: Poor (0), Fair(1), Good(2), Very Good(3), Excellent(4)
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Participants
  Poor | 1 | 4 | 2 | 6 | 15 | 5
  Fair | 6 | 7 | 5 | 4 | 7 | 5
  Good | 7 | 7 | 4 | 7 | 5 | 4
  Very good | 11 | 4 | 9 | 9 | 0 | 11
  Excellent | 2 | 5 | 7 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.35, Cochran-Mantel-Haenszel

22. Secondary Outcome: Number of Times Participants Took Rescue Medication
Description: Subjects were allowed to "rescue" and take a non-study pain reliever if the pain was not tolerable. This measure represents for the number of times rescue medication was taken by a subject.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Participants
  0 | 15 | 15 | 19 | 14 | 2 | 16
  1 | 12 | 12 | 8 | 13 | 22 | 11
  2 | 0 | 0 | 0 | 0 | 3 | 0
  3 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Total Wake Time Measured by Actigraphy
Description: Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Minutes | 253.72 [174 to 333] | 290.03 [210 to 370] | 180.21 [100 to 260] | 285.62 [206 to 365] | 518.58 [439 to 598] | 255.20 [175 to 336]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.53, ANCOVA

24. Secondary Outcome: Sleep Efficiency Measured by Actigraphy
Description: Sleep efficiency was calculated as (total sleep time/total time in-bed time) × 100; total in-bed time was fixed at 10 hours. Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of sleep time
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Percentage of sleep time | 57.24 [44 to 71] | 51.49 [38 to 65] | 68.87 [55 to 82] | 52.09 [39 to 66] | 12.85 [-1 to 26] | 56.70 [43 to 70]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.55, ANCOVA

25. Secondary Outcome: Activity Mean Measured by Actigraphy
Description: Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects. Activity mean - average movement per minute.
Time Frame: Up to 10 hours
Population: ITT (Intent to Treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Movement per minute
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Movement per minute | 42.09 [25 to 59] | 48.48 [32 to 65] | 26.73 [10 to 43] | 52.36 [36 to 69] | 72.43 [56 to 89] | 41.14 [24 to 58]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.59, ANCOVA

26. Secondary Outcome: Wake Episode Measured by Actigraphy
Description: Actigraphy is a non-intrusive tool that measures an individual's movement during sleep. Actigraphy was used to obtain data in discriminating between sleep and wake states in the subjects. Wake Episodes - # of blocks of continuous wake epochs (defined as 2 or more consecutive epochs scored as wake that ends when there is at least one epoch scored as sleep subsequent to the start of the wake epochs).
Time Frame: Up to 10 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: Wake episodes
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
Wake episodes | 8.38 [5 to 11] | 10.86 [8 to 14] | 13.26 [10 to 16] | 9.89 [7 to 13] | 5.84 [3 to 9] | 11.98 [9 to 15]
Statistical Analysis 1: Comparison: Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg vs Naproxen Sodium 440 mg (BAYH6689); Test type: Superiority or Other; p = 0.25, ANCOVA

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected after the administration of the first dose of study drug up to 5 days post drug administration, or up to 30 days after the last study drug administration if they were serious adverse events (SAEs).
Arm/Group | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 440 mg (BAYH6689) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg | Naproxen Sodium 220 mg (BAYH6689) | DPH 50mg | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 2/27 | 2/27 | 3/27 | 1/27 | 5/27 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naproxen Sodium 440 mg (BAYH6689) / DPH 50mg (N=27) | Naproxen Sodium 440 mg (BAYH6689) (N=27) | Naproxen Sodium 220 mg (BAYH6689) / DPH 50mg (N=27) | Naproxen Sodium 220 mg (BAYH6689) (N=27) | DPH 50mg (N=27) | Ibuprofen 400 mg / Diphenhydramine Citrate 76 mg (N=27)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No